CLINICAL TRIAL: NCT01813487
Title: Study of the Immunogenicity and Efficacy of HBsAg Vaccine in Combination With Standard Antiviral Therapy in Patients Who Have Been Treated With HB110E Hepatitis B DNA Vaccine
Brief Title: Study of the Immunogenicity and Efficacy of HBsAg Vaccine in Combination With Standard Antiviral Therapy With HB110E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB110E_PI_PS
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HBsAg vaccine with Entecavir (Other)
  Interventions: Drug: HBsAg vaccine with Entecavir

INTERVENTIONS:
Drug: HBsAg vaccine with Entecavir

SUMMARY:
The purpose of this study is to examine the immunogenicity and efficacy of HBsAg Vaccine in combination with Entecavir in patients who have been treated with HB110E HBV DNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have been treated with HB110E 2mg or 4mg within 6 months prior to screening.
* positive HBsAg at screening
* serum HBV DNA level below 300copies/mL at screening
* ALT level within 2 x ULN at screening
* voluntarily provide the informed consent

Exclusion Criteria:

* participation in other study within 30 days of screening
* subjects with severe allergic reaction or severe adverse event to HBsAg vaccine, or not suitable for HBsAg vaccine.
* any other conditions that are considered inappropriate for the study by the investigator

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: HBV specific T-cell response by ELISPOT | Change from Baseline in HBV specificic T-cell response at 16 weeks
  sample for immunologic assay will be collected at each visit; VS(~4week), VT1(0week), VT2(8week), VF(16week. T-cell response will be measured by ex-vivo & cultured ELISPOT.

SECONDARY OUTCOMES:
HBsAg titer | Change from baseline in HBsAg titer at 16 weeks
  sample for HBsAg will be collected at each visit; VS(~4week), VT1(0week), VT2(8week), VF(16week. Change from baseline in HBsAg titer will be measured at VF.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Yoon, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, South Korea